CLINICAL TRIAL: NCT05139953
Title: Impact of COVID-19 Infection During Pregnancy on Maternal and Fetal Outcome
Brief Title: Impact of COVID-19 Infection During Pregnancy
Status: Completed | Type: Observational
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohamed Elsibai Anter, Assistant professor of obstetrics and gynecology, Menoufia University
Other Study IDs: 4/2021OBSGN18
Record Dates: First submitted 2021-11-29; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Covid-19 in Pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
To asses impact of the COVID-19 infection during Pregnancy on maternal and fetal outcome in relation to gestational age.

DETAILED DESCRIPTION:
COVID-19, caused by SARS-COV-2, was first reported in the city of Wuhan, Hubei province, China, at the end of December 2019. The exact origin of human infection has not yet been clearly identified.SARS-CoV-2 is a member of the Coronavirus family, and other pathogens from this family have inflicted a range of viral infections, including Middle East Respiratory Syndrome (MERS) and Severe Acute Respiratory Syndrome (SARS). The incubation period varies from 2 days to 2 weeks following exposure to the virus.The global pandemic caused by the severe acute respiratory syndrome coronavirus (SARS-CoV-2) has been growing at an accelerating rate. The increasing mortality rate warrants identification and protection of the vulnerable populations in society.It is well known that pregnancy-related immune suppression makes mothers more vulnerable than non-pregnant women to several viral infections, including SARS-COV, hepatitis E virus, influenza, and herpes simplex virus.

Furthermore, changes in pulmonary function during pregnancy, including decreased total lung capacity and functional residual capacity, may cause susceptibility to viral pneumonia.

Data on clinical outcomes of pregnant women suffering from COVID-19 are therefore relatively scarce. Recently a meta-analysis of 13 publications reported preterm births, neonatal pneumonia, and respiratory distress syndrome in infants born of COVID-19-positive mothers. The rates of cesarean deliveries and adverse pregnancy outcomes were substantially higher

ELIGIBILITY:
Inclusion Criteria:

-All medical records of the pregnant women admitted to EL Bagour Quarantine hospital, Menoufia governorate due to SARS-CoV-2 infection, as confirmed by real-time reverse transcriptase-polymerase chain reaction (RT-PCR) assay of nasopharyngeal swab specimens.

Exclusion Criteria:

* Patients who had equivocal or negative testing results were excluded from the study

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: All medical records of pregnant women admitted to EL Bagour Quarantine hospital, Menoufia governorate diagnosed with SARS-CoV-2 infection from May, 2020 were revised to collect maternal and neonatal data using a standardized data collection sheet.
  The Information included:
  * Age
  * GA
  * Parity
  * Pre-existing medical condition
  * Presenting symptoms at admission; such as fever, sore throat/ nasal or sinus congestion, cough/chest pain, vomiting/diarrhea, and fatigue/myalgia, dyspnea….etc.
  * Body mass index.
  * The laboratory results at admission and on discharge
  * Lymphopenia was defined when lymphocytes count less than 1100 cells/mm3.
  * Ultrasound report upon admission to the hospital that included; fetal viability, amniotic fluid index and any placental abnormality.
  * C.T. Report if done.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Studying impact of COVID-19 on pregnancy | baseline
  understanding of the impact of COVID-19 on pregnancy will provide critical data about the course of the disease in pregnant women and their infants .

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed E Anter, MD, Study Director — Menoufia University-Shebin Elkom-Egypt
Locations (1):
- Menoufia University hospital, Shibīn al Kawm, Menoufia, Egypt